CLINICAL TRIAL: NCT03710590
Title: Effects of Electronic Cigarette Settings and Liquid Concentrations in Cigarette Smokers and Electronic Cigarette Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20012738; U54DA036105 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-10-18 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Electronic Cigarettes
MeSH Terms: conditions — Vaping | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to determine differences in nicotine delivery, use behavior (puff topography), carbon monoxide delivery, subjective effects, and physiological effects, when cigarette smokers and experienced electronic cigarette users use an electronic cigarette with different settings (different voltage and resistance settings, which together determine power levels) and different e-liquid concentrations.
Who Masked: Participant
Masking Description: Participants will be blinded to the power level and nicotine concentration used in each session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cigarette smokers (Active Comparator)
  Interventions: Other: ECIG Lab Session 15 watts, 10 mg nicotine; Other: ECIG Lab Session 15 watts, 15 mg nicotine; Other: ECIG Lab Session 15 watts, 30 mg nicotine; Other: ECIG Lab Session 30 watts, 10 mg nicotine; Other: ECIG Lab Session 30 watts, 15 mg nicotine; Other: ECIG Lab Session 30 watts, 30 mg nicotine
- Electronic cigarette users (Active Comparator)
  Interventions: Other: ECIG Lab Session 15 watts, 10 mg nicotine; Other: ECIG Lab Session 15 watts, 15 mg nicotine; Other: ECIG Lab Session 15 watts, 30 mg nicotine; Other: ECIG Lab Session 30 watts, 10 mg nicotine; Other: ECIG Lab Session 30 watts, 15 mg nicotine; Other: ECIG Lab Session 30 watts, 30 mg nicotine

INTERVENTIONS:
Other: ECIG Lab Session 15 watts, 10 mg nicotine — During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Other: ECIG Lab Session 15 watts, 15 mg nicotine — During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.).
Other: ECIG Lab Session 15 watts, 30 mg nicotine — During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Other: ECIG Lab Session 30 watts, 10 mg nicotine — During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Other: ECIG Lab Session 30 watts, 15 mg nicotine — During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
Other: ECIG Lab Session 30 watts, 30 mg nicotine — During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.

SUMMARY:
The purpose of this research study is to find out how different types of electronic cigarettes (ECIG) settings, combined with e-liquids of differing nicotine concentrations, affect blood nicotine levels, use behavior (how users puff), and how users feel.

ELIGIBILITY:
Inclusion Criteria--participants must be:

* healthy (determined by self-report)
* between the ages of 18-55
* willing to provide informed consent
* able to attend the lab and abstain from tobacco/nicotine as required and must agree to use designated products according to study protocol

Exclusion Criteria:

* Women if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.
* Individuals who weigh less than 110 pounds

Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Clinical Behavioral Pharmacolgy Laboratory, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eversole A, Budd S, Karaoghlanian N, Lipato T, Eissenberg T, Breland AB. Interactive effects of protonated nicotine concentration and device power on ENDS nicotine delivery, puff topography, and subjective effects. Exp Clin Psychopharmacol. 2023 Apr;31(2):443-454. doi: 10.1037/pha0000576. Epub 2022 Jun 13. PMID 35696157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Not-completed reason was not stored by treatment arm
Pre-assignment Details: Each participant will participate in 6 sessions. Sessions differ by the tobacco product used (see study arms). The sessions are ordered by latin-square; however, session order was NOT expected to change any outcomes and order effects are not relevant to the study. Therefore all outcome data was merged and analyzed only by arm and session without regard to order.
Groups:
- Cigarette Smokers; E-cigarette Users: Each participant will participate in 6 sessions. During each session, participants will first complete a 10-puff product use bout, and then a 90-minute ad lib product use bout.
  Session 1: ECIG Lab Session 15 watts, 10 mg nicotine Session 2: ECIG Lab Session 15 watts, 15 mg nicotine Session 3: ECIG Lab Session 15 watts, 30 mg nicotine Session 4: ECIG Lab Session 30 watts, 10 mg nicotine Session 5: ECIG Lab Session 30 watts, 15 mg nicotine Session 6: ECIG Lab Session 30 watts, 30 mg nicotine
Period: Overall Study
Arm/Group | Cigarette Smokers | E-cigarette Users
Started | 22 | 23
Session 1: ECIG Lab Session 15 Watts, 10 mg Nicotine | 12 | 15
Session 2: ECIG Lab Session 15 Watts, 15 mg Nicotine | 12 | 15
Session 3: ECIG Lab Session 15 Watts, 30 mg Nicotine | 12 | 15
Session 4: ECIG Lab Session 30 Watts, 10 mg Nicotine | 12 | 15
Session 5: ECIG Lab Session 30 Watts, 15 mg Nicotine | 12 | 15
Session 6: ECIG Lab Session 30 Watts, 30 mg Nicotine | 12 | 15
Completed | 12 | 15
Not Completed | 10 | 8
Not completed — Lost to follow up, study stopped due to COVID-19, other reasons | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cigarette Smokers | E-cigarette Users | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.67 (8.74) | 25.40 (7.94) | 29.07 (9.15)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 7 | 8 | 15
  Other | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 7 | 11 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Nicotine
Description: Change in plasma nicotine level.
Time Frame: Baseline to 5 min after the start of a 10-puff product use
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cigarette Smokers | E-cigarette Users
Number analyzed (Participants) | 12 | 15
ng/ml
  10mg 15 Watts | 8.68 (7.22) | 8.28 (9.65)
  10mg 30 Watts | 9.53 (7.53) | 12.00 (10.29)
  15mg 15 Watts | 7.34 (6.19) | 7.17 (6.14)
  15mg 30 Watts | 13.04 (13.14) | 14.04 (12.08)
  30mg 15 Watts | 10.18 (9.28) | 20.12 (22.40)
  30mg 30 Watts | 17.28 (18.05) | 22.38 (21.04)

2. Primary Outcome: Puff Volume
Description: The average volume of each puff, in ml, during 10 puff bout.
Time Frame: Each time the e-cigarette is used during the 10-puff use bout - 5 minutes
Population: One participant did not have data for this measure.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Cigarette Smokers | E-cigarette Users
Number analyzed (Participants) | 11 | 15
ml
  10 mg, 15 Watts | 457.27 (223.02) | 748.34 (412.22)
  10 mg, 30 Watts | 245.11 (124.09) | 503.43 (216.28)
  15 mg, 15 Watts | 350.18 (190.97) | 708.62 (300.45)
  15 mg, 30 Watts | 217.01 (94.99) | 409.56 (208.61)
  30 mg, 15 Watts | 310.95 (199.06) | 631.23 (225.84)
  30 mg, 30 Watts | 176.32 (79.76) | 415.85 (186.33)

3. Primary Outcome: Puff Duration
Description: The average duration of each puff, in seconds.
Time Frame: Each time the e-cigarette is used during the 10-puff use bout - 5 minutes
Population: One participant did not have data collected for this measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cigarette Smokers | E-cigarette Users
Number analyzed (Participants) | 11 | 15
seconds
  10 mg, 15 W | 3.04 (1.01) | 4.37 (1.15)
  10 mg, 30 W | 1.97 (0.65) | 2.83 (0.71)
  15 mg, 15 W | 2.59 (0.53) | 4.02 (1.27)
  15 mg, 30 W | 1.65 (0.43) | 2.72 (1.05)
  30 mg, 15 W | 2.44 (0.83) | 3.41 (1.01)
  30 mg, 30 W | 1.58 (0.45) | 2.45 (0.84)

4. Secondary Outcome: Heart Rate
Description: Average heart rate, measured in beats per minute.
Time Frame: Heart rate will be measured from baseline continuously throughout the 10-puff bout - 5 minutes
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cigarette Smokers | E-cigarette Users
Number analyzed (Participants) | 12 | 15
bpm
  10 mg, 15 Watts | 75.66 (6.88) | 75.01 (10.44)
  10 mg, 30 Watts | 78.19 (7.25) | 79.92 (15.30)
  15 mg, 15 Watts | 72.64 (6.32) | 79.09 (15.30)
  15 mg, 30 Watts | 76.05 (6.91) | 80.27 (12.51)
  30 mg, 15 Watts | 77.12 (8.83) | 78.56 (12.67)
  30 mg, 30 Watts | 80.12 (8.95) | 84.51 (14.79)

5. Other Pre Specified Outcome: Inter Puff Interval
Description: The time between each puff, in seconds
Time Frame: Inter puff interval will be measured each time the e-cigarette is used during an approximately 4 hour session: during a 5-minute 10-puff use bout, and during an approximately 90 minute ad lib use period
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Flow Rate
Description: The rate of air flow during each puff, in ml/second
Time Frame: Flow rate will be measured each time the e-cigarette is used during an approximately 4 hour session: during a 5-minute 10-puff use bout, and during an approximately 90 minute ad lib use period
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Hughes-Hatsukami Questionnaire
Description: This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 11 items scored 0 - 100, with lower scores indicating less severe symptoms. There are no sub-scales. Items are analyzed separately.
Time Frame: Questionnaire will be administered 4 times in each each approximately 4-hr session: before any product use, 10 minutes after the start of a 10-puff use bout, and then before and after an approximately 1-hour ad lib use period.
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Direct Effects of Product Use Questionnaire
Description: This scale is used to assess how product use makes participants feel and consists of 10 questions that are scored 0 - 100. There are no sub-scales. Items are analyzed separately.
Time Frame: Questionnaire will be administered 2 times in each each approximately 4-hr session: 10 minutes after the start of a 10-puff use bout, and then after an approximately 1-hour ad lib use period.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Direct Effects of Nicotine Questionnaire
Description: This scale is used to assess how product use makes participants feel, and consists of 10 questions that are scored 0 - 100.There are no sub-scales. Items are analyzed separately.
Time Frame: as for outcome 7
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Carbon Monoxide Levels
Description: Change in carbon monoxide levels (in parts per mission)
Time Frame: Carbon monoxide levels will be assessed before and after product use in each approximately 4-hr session: at baseline, 5 min after the end of a 10-puff product use, and then before and after an approximately 1-hour ad lib use period.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Blood Pressure
Description: Change in blood pressure, measured in mm/hg
Time Frame: Blood pressure will be measured from baseline continuously throughout each approximately 4-hr session
Reporting Status: Not Posted

12. Other Pre Specified Outcome: General Labeled Magnitude Scale
Description: This scale measures the flavor sensation, harshness, and throat hit (in three questions that correspond to those constructs) of the e-cigarette used in each session. The scale ranges from 0 - 100, with 0 being no sensation and 100 being the strongest imaginable sensation of any kind. Each item if scored nd analyzed separately (there are no sub-scales).
Time Frame: The General Labeled Magnitude Scale will be administered twice in each approximately 4 hour session--after a 5-minute 10 puff use bout, and after the approximately 90 minute ad lib period.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During each of 6 approximately 4-hour session over up to a 3 week period.
Description: This study did not have any SAEs or all-cause mortality.
Arm/Group | Cigarette Smokers | E-cigarette Users
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT03710590/Prot_SAP_001.pdf
  • Informed Consent Form (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT03710590/ICF_000.pdf